CLINICAL TRIAL: NCT04988906
Title: Monitoring Ventilations During Out-of-Hospital Cardiac Arrest Resuscitation
Brief Title: Ventilation Monitoring in OHCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Prescott-Russell Paramedic Service (Unknown); Peterborough Paramedic Service (Unknown); Bruce County Paramedic Service (Unknown); Waterloo Paramedic Service (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 1987
Record Dates: First submitted 2021-07-16; First posted 2021-08-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Ventilation; Cardiac Arrest; Resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Respiratory Aspiration; Heart Arrest

STUDY DESIGN:
Intervention Model Description: Before-and-After Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before Arm (No Intervention): The before arm of the study prehospital providers will provide resuscitation as per standard practice. The providers will utilize the Zoll Accuvent device without activation of the real-time dashboard. This will allow us to collect baseline ventilation data.
- After Arm (Active Comparator): The after arm of the study the prehospital providers will provide resuscitation as per standard practice. The real-time ventilation dashboard will be activated and the providers will use real-time feedback to monitor ventilation quality during the resuscitation.
  Interventions: Device: Zoll Accuvent Ventilation Monitor

INTERVENTIONS:
Device: Zoll Accuvent Ventilation Monitor — Provides real-time ventilation quality monitoring (rate and volume)
  Arms: After Arm

SUMMARY:
This is a before-and-after study examining the impact of real-time ventilation monitoring during out-of-hospital cardiac arrest. Study investigators will compare ventilation quality (rate, volume) performed during the resuscitation without the real-time feedback (before phase), to ventilation quality with the use of real-time feedback using the Zoll Accuvent device (after phase).

DETAILED DESCRIPTION:
The before intervention phase of this study will involve no change in practice to cardiac resuscitation by paramedics. Paramedics will be instructed to attach the Zoll AccuVent® to the BVM at each use and to leave it attached throughout the duration of the resuscitation.

During the resuscitation the Zoll AccuVent® will monitor and record ventilation rates and volumes that are being delivered during each ventilation performed utilizing the "Real BVM Help®" dashboard, however rescuers will be blinded to this information and will not be able to access it during the resuscitation. Post-call paramedics will upload the Zoll file containing the ventilation data in addition to CPR quality data and cardiac rhythms. This is consistent with current standard practice. These files will then be used by study investigators for data analysis. During this initial phase, to avoid biasing the study results the paramedics will only be trained on application of the Zoll AccuVent®, but will not have access to the real-time dashboard.

The study intervention will involve a brief training session for paramedics during the annual continuing medical education (CME) day. Training will consist of specifics of the study as well as how to apply the Zoll AccuVent® device and use the device during a cardiac arrest. Paramedics will be reminded of good ventilation practices during cardiac arrest and post-cardiac arrest care as well as current standards of practice as defined by the American Heart Association and Heart and Stroke Foundation of Canada.

Post-intervention, paramedics will be "un-blinded" and able to utilize the real-time feedback from the Zoll AccuVent® to help guide the delivery of ventilations during cardiac arrest resuscitation. All other aspects of care will be provided in accordance with standard practice at that time. Once the Zoll AccuVent® is applied, paramedics will use the real-time monitoring capabilities of the device to monitor the delivery of ventilations (rate and volume) during the resuscitation. Post-call paramedics will again upload files containing ventilation data that study investigators will analyze to compare our results.

Bivariate descriptive statistics will be used to examine differences in ventilation parameters between paramedics while using the Zoll AccuVent® and using standard monitoring devices (standard of care). The mean volume (mL) will be calculated for each of the two groups and Student's t-test will be used to compare the mean difference in volume (mL) between groups. Investigators will compare the proportion of ventilations per minute that are compliant with AHA guideline recommendations using Chi-square test for proportions.

The relationship between ventilations (volume and rate) and ROSC will be assessed using Poisson regression with robust standard errors. The results will be reported as relative risks (RR) and 95% confidence intervals for each of the included variables.

The volume of ventilations (mL) will be evaluated as a continuous variable, with secondary analyses analyzing per increase of 10mL as well as by quintiles of ventilation volume provided. The rate of ventilations will be analyzed categorically as "Compliant (8-10 per minute)", "Too Slow (< 8 per minute)", or "Too Fast (> 10 per minute)". Regression models will control for standard Utstein variables and additional modelling will examine for interactions between ventilation parameters and patient sex, patient age, initial rhythm and witness status. If a significant interaction is found subgroup analyses will be performed examining these specific groups.

A priori subgroup analyses will be performed examining differences between airway strategies (BVM vs. endotracheal intubation vs. supraglottic airway) as well as intra-arrest and post-arrest management.

ELIGIBILITY:
Inclusion Criteria:

* All adult out-of-hospital cardiac arrests treated by paramedics

Exclusion Criteria:

* traumatic cardiac arrest
* prehospital Do Not Resuscitate (DNR) orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Ventilation Volume | Day 1
  Measurement of the volume of ventilation (mL) during resuscitation

SECONDARY OUTCOMES:
Feasibility of successfully using Zoll Accuvent device in the field Feasibility | Day 1
  Ability to use the Zoll Accuvent during the resuscitation, obtain feedback, and download ventilation information. Feasibility will be defined as >80% success rate.
Prehospital Return of spontaneous circulation (ROSC) | Day 1
  any return of circulation in the prehospital setting as documented by paramedics
Ventilation Rate | Day 1
  Measure the rate (per minute) of ventilations delivered during resuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No